CLINICAL TRIAL: NCT04259346
Title: Bioequivalence of an Alternate Ixekizumab Formulation Compared to the Commercial Formulation in Healthy Subjects
Brief Title: A Study of Two Formulations of Ixekizumab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17151; I1F-MC-RHCU (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-02-01

CONDITIONS: Healthy
MeSH Terms: interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ixekizumab (Reference) (Experimental): Approved formulation of 80 milligram (mg) ixekizumab administered as a subcutaneous (SC) injection via autoinjector (AI).
  Interventions: Drug: Ixekizumab
- Ixekizumab (Test) (Experimental): Test formulation of 80 mg ixekizumab administered as a SC injection via AI.
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Ixekizumab — Administered SC.
  Other Names: LY2439821

SUMMARY:
The purpose of this study is to compare two different formulations of ixekizumab. One formulation (Reference) is approved by the Food and Drug Administration (FDA) and one formulation (Test) is not approved. This study will compare how much of each formulation gets into the blood stream. Information about any side effects that may occur will also be collected. The study will last up to about four months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy male or female participants, with chronic stable medical problems, that in the investigator's opinion will not place the subject at increased risk by participating in the study

Exclusion Criteria:

* Have a significant history of, or current, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or hematologic disorders that in the opinion of the investigator poses an unacceptable risk to the participant if participating in the study
* Are allergic or hypersensitive to the study medicine
* Had a vaccination with a live vaccine within 12 months prior to the first check-in or intend to get a vaccine for tuberculosis within 12 months of completing treatment on this study
* Have any type of hepatitis, human immunodeficiency virus (HIV) infection, or other serious infection
* Show evidence of active or latent tuberculosis (TB)
* Presence of significant neuropsychiatric disorder or a recent history of depression
* Have had any active or recent infection within 4 weeks of Day 1 that, in the opinion of the investigator, would pose an unacceptable risk to the participant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - Miami Research Associates, Miami, Florida
  - Covance Dallas, Dallas, Texas
  - Covance Clinical Research Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chabra S, Gill BJ, Gallo G, Zhu D, Pitou C, Payne CD, Accioly A, Puig L. Ixekizumab Citrate-Free Formulation: Results from Two Clinical Trials. Adv Ther. 2022 Jun;39(6):2862-2872. doi: 10.1007/s12325-022-02126-0. Epub 2022 Apr 21. PMID 35449322

RESULTS

PARTICIPANT FLOW:
Groups:
- 80 Milligram (mg) Ixekizumab (Reference): Participants received 80 mg ixekizumab of approved commercial formulation (Reference) administered as a subcutaneous (SC) injection via autoinjector (AI).
- 80 mg Ixekizumab (Test): Participants received 80 mg ixekizumab alternate formulation (Test) administered as a SC injection via AI.
Period: Overall Study
Arm/Group | 80 Milligram (mg) Ixekizumab (Reference) | 80 mg Ixekizumab (Test)
Started | 126 | 119
Received at Least One Dose of Study Drug | 126 | 119
Completed | 122 | 115
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 80 mg Ixekizumab (Reference): Participants received 80 mg ixekizumab of approved commercial formulation (Reference) administered as a SC injection via AI.
- Total: Total of all reporting groups
Arm/Group | 80 mg Ixekizumab (Reference) | 80 mg Ixekizumab (Test) | Total
Number analyzed (Participants) | 126 | 119 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (12.8) | 46.8 (13.5) | 44.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 60 | 127
  Male | 59 | 59 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 46 | 104
  Not Hispanic or Latino | 68 | 73 | 141
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 19 | 51
  White | 93 | 98 | 191
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 126 | 119 | 245

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Ixekizumab
Description: PK: Cmax of ixekizumab was evaluated
Time Frame: Predose, Day 3, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 Post Dose
Population: Only participants who had all PK samples collected up to Day 85 or participants who had one missing PK sample after Day 15 but with at least 3 data points and R squared adjusted (Rsq adj) greater than (>) 0.7 to calculate half-life parameter included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | 80 mg Ixekizumab (Reference) | 80 mg Ixekizumab (Test)
Number analyzed (Participants) | 112 | 110
micrograms per milliliter (ug/mL) | 9.66 (33) | 9.97 (35)

2. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Ixekizumab
Description: Area under the plasma concentration versus time curve from time zero to the last measured concentration value (AUC[0-tlast]). AUC 0-tlast is equal to AUC (0-85) days where the last time point was 85 Days ± 3 Days.
Time Frame: Predose, Day 3, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 Post Dose
Population: Only participants who had all PK samples collected up to Day 85 or participants who had one missing PK sample after Day 15 but with at least 3 data points and Rsq adj>0.7 to calculate half-life parameter included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day/milliliter (ug*day/mL)
Arm/Group | 80 mg Ixekizumab (Reference) | 80 mg Ixekizumab (Test)
Number analyzed (Participants) | 112 | 110
microgram*day/milliliter (ug*day/mL) | 207 (31) | 219 (28)

3. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Ixekizumab
Description: Area under the plasma concentration versus time curve from zero to infinity (AUC[0-∞]) of a single dose of Ixekizumab.
Time Frame: Predose, Day 3, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 Post Dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*day/mL
Arm/Group | 80 mg Ixekizumab (Reference) | 80 mg Ixekizumab (Test)
Number analyzed (Participants) | 112 | 110
ug*day/mL | 213 (33) | 227 (30)

ADVERSE EVENTS:
Time Frame: Up to 85 Days
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 80 mg Ixekizumab (Reference) | 80 mg Ixekizumab (Test)
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/119
Other Adverse Events (participants affected / at risk) | 36/126 | 14/119
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mg Ixekizumab (Reference) (N=126) | 80 mg Ixekizumab (Test) (N=119)
Injection site reaction (General disorders) | 30 (30) | 11 (11)
Headache (Nervous system disorders) | 9 (11) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT04259346/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT04259346/SAP_001.pdf